CLINICAL TRIAL: NCT05448326
Title: The Diagnostic Observatory: Combating Diagnostic Wandering and Impasse Within the AnDDI-Rares Network
Acronym: Obs du Diag
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE 2021
Record Dates: First submitted 2022-06-01; First posted 2022-07-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Developmental Abnormality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Work package 1 (WP1): Patients without a diagnosis who consulted for a developmental anomaly in 2012 and 2022 and agree to resume a diagnostic approach
  Interventions: Other: Questionnaire to assess expectations of a diagnosis
- Work package 2 (WP2): Part 1 (Lab): Patients with developmental abnormalities with or without neurodevelopmental disorders who have had a CNV (Copy Number Variation) rendering that remained of unknown significance or classified as (probably) benign Part 2 (Clinical part): Patients who agree to resume the diagnostic process following a CNV report of unknown significance or classified as (probably) benign
  Interventions: Other: Questionnaire to assess understanding of previously reported results and expectations of a diagnosis
- Work package 3 (WP3): Patients with an established clinical diagnosis belonging to the characteristic syndromes of the AnDDI-Rares network (known gene(s) but negative molecular diagnosis)
  Interventions: Biological: Blood sample +/- skin biopsy

INTERVENTIONS:
Other: Questionnaire to assess expectations of a diagnosis — Duration 45 minutes
  Groups: Work package 1 (WP1)
Other: Questionnaire to assess understanding of previously reported results and expectations of a diagnosis — Duration 30 minutes
  Groups: Work package 2 (WP2)
Biological: Blood sample +/- skin biopsy — 8 ml of blood biopsy: size 3 to 5 mm
  Groups: Work package 3 (WP3)

SUMMARY:
The Direction Générale de l'Organisation des Soins (DGOS) and the Banque Nationale de Données Maladies Rares (BNDMR) have launched a call for a letter of commitment for the implementation of a diagnostic observatory in order to fight against diagnostic wandering and impasse. In this context, the AnDDI-Rares network proposes 3 work packages (WP) to respond to the missions entrusted to it.

Work package 1 of the diagnostic observatory includes a retrospective and prospective study to evaluate how diagnostic wandering and impasse has evolved within the network, with regard to the integration of new technologies, and the expectations of patients and their families.

Work package 2 of the diagnostic observatory includes a reassessment of sporadic copy number variations (CNV) of unknown significance of more than 1 Mb obtained since the beginning of CGH array analyses in the territory.

Work package 3 of the diagnostic observatory aims to help put an end to diagnostic wandering for patients with certain emblematic syndromes by proposing genome and RNA analysis, which provides a certain diagnosis and negative targeted molecular study.

ELIGIBILITY:
Inclusion Criteria:

WP1:

- Children or adult patients who did not obtain a diagnosis after consulting for a developmental abnormality (that may include isolated or multiple, minor or major malformations, facial dysmorphia associated or not with learning disabilities and/or intellectual disability). These patients had a diagnostic evaluation over the 2 weeks randomly drawn from 2012 and 2022.

Patients agreeing to resume a diagnostic approach requiring new blood samples. For genome sequencing through the platforms of the France Genomic Medicine Plan, when they correspond to the criteria of existing preindications, the parents' sample will be proposed.

- Patients (adults or their parents) affiliated to national health insurance or beneficiaries of such a system

WP2:

For the identification of patients eligible for reanalysis (Part 1 Lab) :

* Patients, children or adults with developmental anomalies with or without neurodevelopmental disorders,
* Patients in whim a de novo CNV of unknown significance of more than 1 Mb has been detected since the implementation of the CGH array platforms
* The CNV remained of unknown significance or classified as (probably) benign after reanalysis* *reanalysis other than that performed in the context of the diagnostic observatory

For reanalysis, in addition to the previous inclusion criteria (Part 2 Clinical):

* CNV remained of unknown significance or classified as (probably) benign after reanalysis**
* Patients and/or their parents agreeing to resume diagnostic testing
* Patients (adults or their parents) affiliated to national health insurance or beneficiaries of such a system ** After reanalysis in the framework of the diagnostic observatory

WP3:

* Patients (children or adults) with a syndrome that corresponds to the study criteria:
* Established clinical diagnosis for one of the characteristic syndromes of the AnDDI-Rares pipeline (list may be revised in the future): Noonan syndrome, CHARGE syndrome, Kabuki syndrome, Cornelia de Lange syndrome, Rubinstein-Taybi syndrome ;
* Known gene(s) but patient's molecular diagnosis is negative.
* Patients and at least one parent agreeing to a new blood sample for genome ± RNA sequencing and/or skin biopsy for conditions where gene transcription is not satisfactory from RNA extracted from blood; or agreeing to perform these analyses from previously stored samples (recommended trio - trio may include other family members);
* Parents of legal age who are affiliated with national health insurance or who are beneficiaries of such a system;
* Signed informed consent from both biological parents and/or the index case if they are of legal age;
* Ability of both biological parents to understand correctly.

Exclusion Criteria:

WP1:

* Patients without a developmental abnormality ;
* Patients with a previously identified diagnosis at the time of consultations on the weeks drawn randomly from 2012 and 2022.

WP3:

* Unlikely clinical diagnosis ;
* Family not wishing to pursue molecular investigations;
* Index case having already benefited from the investigations through another research project.
* The parents of the index case are under court protection ;
* Families where both parental authority holders are not the biological parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in a situation of diagnostic wandering or impasse
Sampling Method: Non-Probability Sample
Enrollment: 1280 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Consultations leading to a causal genetic diagnosis in 2012 and 2022 | through study completion, an average of 24 months
CNVs reclassified as pathogenic/probably pathogenic or benign/probably benign. | through study completion, an average of 24 months
Molecular diagnosis identified by sequencing of the genome ± associated RNA. | through study completion, an average of 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France